CLINICAL TRIAL: NCT03613038
Title: Understanding Communication and Cognitive Impairments in Neurodegenerative Disorders
Brief Title: A Systematic Investigation of Phonetic Complexity Effects on Articulatory Motor Performance in Progressive Dysarthria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Mili Kuruvilla, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1209643; 1R15DC016383-01 (NIH)
Record Dates: First submitted 2018-07-10; First posted 2018-08-02 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Amyotrophic Lateral Sclerosis; Parkinson Disease
Keywords: Dysarthria; Speech motor performance; Speech motor control; Speech kinematics
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Parkinson Disease; Dysarthria

STUDY DESIGN:
Intervention Model Description: Two groups of participants i.e., participants with ALS or PD and healthy controls will be asked to repeat sentences that have target words with varying phonetic complexity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phonetic complexity effects (Other): Conduct a comprehensive kinematic assessment using state-of-the art 3D speech tracking technology on individuals with ALS and PD as well as healthy talkers to identify articulatory motor disturbances as a function of phonetic complexity and dysarthria severity. Phonetic complexity will be experimentally manipulated using the consonant and vowel complexity classification system proposed by Kent (1992) that takes into account the underlying articulatory motor adjustments required to produce various speech sounds.
  Interventions: Behavioral: Phonetic complexity effects on speech motor performance

INTERVENTIONS:
Behavioral: Phonetic complexity effects on speech motor performance — Use of 3D electromagnetic articulography to examine phonetic complexity effects of single word stimuli at the articulatory kinematic level in talkers each with preclinical, mild, and moderate dysarthria, relative to healthy controls.

SUMMARY:
The goal is to improve the fundamental knowledge about articulatory motor performance in people with Lou Gehrig's disease (also known as ALS) and Parkinson's disease (PD), in order to develop more sensitive assessments for progressive speech loss, which may lead to the improved timing of speech therapies.

DETAILED DESCRIPTION:
The long-term goal is to optimize dysarthria assessment by improving the early detection and tracking of articulatory performance in progressive dysarthrias. The short-term goal of the proposed cross-sectional study is to focus on ALS and PD and quantify articulatory kinematic performance as a function of phonetic complexity, which is experimentally manipulated based on theoretical principles of speech motor development. The research strategy is to use 3D electromagnetic articulography to examine phonetic complexity effects of single word stimuli at the articulatory kinematic level in 15 talkers each with preclinical, mild, and moderate dysarthria, relative to 45 controls. The central hypothesis is that as dysarthria severity increases the discrepancy in articulatory performance, indexed by movement speed, distance, coordination, and variability, between people with dysarthria and typical controls will significantly increase at a lower phonetic complexity level.

ELIGIBILITY:
Inclusion Criteria:

1. May or may not have a neurological impairment.
2. Age range of 19-90 years.
3. Male or female.
4. Provide written consent before any study specific procedures are performed.
5. Have ability to comply with basic instructions.
6. Monolingual English speaker.
7. Have ability to partake in a 90 minute data collection.

Exclusion Criteria:

1. Any speech, language, cognition, or hearing impairment prior to diagnosis of a neurodegenerative disease.
2. Anyone not appropriate for study participation, as deemed by the principal investigator.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Peak movement speed | Up to 3 months after enrollment
  Peak speed (millimeters/second) for each articulatory marker is the maximum value of the first-order derivative of each marker's Euclidean distance time-history.
Range of movement | Up to 3 months after enrollment
  The convex hull represents the smallest convex set containing all the points in the 3D motion path.
Duration | Up to 3 months after enrollment
  Word duration (seconds) is the time between onset and offset of movement for each word.
Spatiotemporal movement variability (STI) | Up to 3 months after enrollment
  STI is the most widely used metric to capture movement pattern variability during speech. To determine STI, the pattern of articulatory movements and the variability of that pattern over several repetitions of an utterance are examined.
Inter-articulator coordination | Up to 3 months after enrollment
  Spatiotemporal coupling relations between articulators will be derived from vertical movements of the articulators using a covariance measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mili Kuruvilla-Dugdale, PhD, Principal Investigator — University of Missouri-Columbia
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Fairway, Kansas
  - University of Missouri-Columbia, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: Yes
The data collected during this study, especially from people with ALS, cannot be easily duplicated so it will be readily shared with other researchers conducting motor speech research. In addition, few investigators have access to tongue tracking technology; therefore, making the tongue kinematic data available will allow other investigators to answer pertinent questions related to speech decline in progressive dysarthrias. Both the raw data and processed data will be made available to interested investigators but will be devoid of identifiers in order to protect the privacy of the participants. Data documentation such as descriptors and units will also be shared to prevent misinterpretation or confusion. Besides the data itself, the PI is willing to share the stimuli as requested by other investigators.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be ensured as soon as the study starts and even after the study ends.
Access Criteria: Data will only be shared for research purposes.